CLINICAL TRIAL: NCT03398057
Title: Effect of Health Education on Female Teachers' Knowledge and Practices Regarding Early Breast Cancer Detection and Screening in the Jazan Area: A Quasi-Experimental Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anwar Ali Ahmad Alameer (Other Government)
Responsible Party: Sponsor-Investigator, Anwar Ali Ahmad Alameer, R4 physician in community medicine residency program in southern region. Principal investigator. Jazan Health Directorate, Ministry of Health, Jazan, Saudi Arabia, Saudi Commission for Health Specialties, Saudi Arabia
Organization: Saudi Commission for Health Specialties, Saudi Arabia (Other Government)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AAAAlameer
Record Dates: First submitted 2017-12-28; First posted 2018-01-12 (Actual); Last update posted 2018-05-07 (Actual); Status verified 2018-05

CONDITIONS: Effect of Health Education Regarding Screening Tools of Breast Cancer
Keywords: Breast cancer screening; health education; breast self-examination; clinical breast examination; mammography.
MeSH Terms: conditions — Health Education; Breast Self-Examination | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Health education group(intervention group) (Experimental): Standardized heath education Program(SHEP) applied to this group participants .
  Interventions: Other: Health education
- Control group (Placebo Comparator): Placebo health education.
  Interventions: Other: Control group

INTERVENTIONS:
Other: Health education — SHEP included a comprehensive lecture about BC, with a generally deep focus on detection and screening tools, which were illustrated by a PowerPoint presentation with pictures and videos. The program also included a practical session about BSE (on breast silicon model). At the end of SHEP, a focused group discussion was conducted to answer participants' questions, and to discuss important barriers regarding BSE practice and visiting primary health care centers or clinics to undergo CBE and mammography. Different scientific and administrative solutions were discussed. SHEP materials were distributed as a hard copy (booklet) and in electronic format (CD) for all participants in the health education group at the end of training.
  Arms: Health education group(intervention group)
Other: Control group — Placebo health education (pamphlets) will be applied to this group participants during study.
  Arms: Control group

SUMMARY:
The purpose of this study is to assess the effectiveness of health education in improving the knowledge and practices of female teachers regarding screening tools and the early detection of breast cancer.

DETAILED DESCRIPTION:
A two-group quasi-experimental design was conducted among 150 female teachers, who were selected from 75 schools of the Jazan General Administration of Education. Schools were chosen by a simple cluster randomization method. Schools were non-randomly assigned to either the intervention or control group. Eligible participants were recruited by a simple randomization method, proportional to the total number of teachers at each school. Those in the intervention group (n=75 teachers) were compared to the control group (n=75 teachers) at baseline, as well as at 6 weeks and 3 months post-intervention.

Study aim:

Assess effectiveness of health education on improving knowledge and practices regarding Breast cancer(BC) early detection and screening tools among female teachers after six weeks, three months in health education group in compare with control group.

Specific objectives:

Estimate level of awareness among female teachers regarding knowledge and practices of BC early detection and screening tools in Jazan area schools.

Measure the impact of health education on female teachers knowledge and practices regarding BC early detection and screening tools in health education group in compare with control group. So Research questions are:

What is the current awareness level of female teachers in Jazan area schools regarding knowledge and practices of BC early detection and screening tools? Does health education improve knowledge and practices regarding BC early detection and screening tools among female teachers in Jazan area schools in health education group more than control group?

ELIGIBILITY:
Inclusion Criteria:

* 20 years. No personal history of BC. No first degree relative of BC. Not being pregnant or breast feeding. Ability to understand questionnaire

Exclusion Criteria:

Refused to give informed consent. Sever medical problem prevent participation.

Min Age: 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — ≥ 20 years. No personal history of BC. No first degree relative of BC. Not being pregnant or breast feeding. Ability to understand questionnaire
Enrollment: 150 (Actual)
Dates: Start 2017-11-20 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-03-15 (Actual)

PRIMARY OUTCOMES:
Effectiveness of health education on improving knowledge and practice regarding BC screening tools in health education group(75 female teachers) VS control group(75 female teachers) | Researchers assessed the improvement of participants knowledge and practice six weeks after applying of health education programs in both groups.
  Researchers assessed knowledge regarding BC detection and screening tools,through modified version of BCK test questionnaire which originally developed by Kathryn L.McCance,1989, USA, it contains nineteen questions. BSE knowledge and practices were assessed through BSE scale which developed by Champion,V.L.,1984, it contains fifteen questions.
  Researchers assessed clinical breast examination (CBE) and mammography practice through questions from ''Detection of Breast Cancer: Knowledge, Attitude, and Practice of Family Health Strategy Women'' questionnaire by de Oliveria RD and ''Intervention Tailoring for Chinese American Women: Comparing the Effect of Two Video on Knowledge, Attitudes, Intentions to Obtain a Mammogram'' questionnaire by Wang JH, it contains 4 questions.All previous questionnaires are valid and reliable instruments.
Effectiveness of health education on improving knowledge and practice regarding BC screening tools in health education group(75 female teachers) VS control group(75 female | Researchers assessed the improvement of participants knowledge and practice three months after applying of health education programs in both groups.
  Researchers assessed knowledge regarding BC detection and screening tools,through modified version of BCK test questionnaire which originally developed by Kathryn L.McCance,1989, USA, it contains nineteen questions. BSE knowledge and practices were assessed through BSE scale which developed by Champion,V.L.,1984, it contains fifteen questions.
  Researchers assessed clinical breast examination (CBE) and mammography practice through questions from ''Detection of Breast Cancer: Knowledge, Attitude, and Practice of Family Health Strategy Women'' questionnaire by de Oliveria RD and ''Intervention Tailoring for Chinese American Women: Comparing the Effect of Two Video on Knowledge, Attitudes, Intentions to Obtain a Mammogram'' questionnaire by Wang JH, it contains 4 questions.All previous questionnaires are valid and reliable instruments.

SECONDARY OUTCOMES:
Baseline knowledge and practice regarding BC screening tools in health education group(75 female teachers) VS control group(75 female teachers) | At the beginning of study, before applying of health education in both groups
  Researchers assessed knowledge regarding BC detection and screening tools,through modified version of BCK test questionnaire which originally developed by Kathryn L.McCance,1989, USA, it contains nineteen questions. BSE knowledge and practices were assessed through BSE scale which developed by Champion,V.L.,1984, it contains fifteen questions.
  Researchers assessed clinical breast examination (CBE) and mammography practice through questions from ''Detection of Breast Cancer: Knowledge, Attitude, and Practice of Family Health Strategy Women'' questionnaire by de Oliveria RD and ''Intervention Tailoring for Chinese American Women: Comparing the Effect of Two Video on Knowledge, Attitudes, Intentions to Obtain a Mammogram'' questionnaire by Wang JH, it contains 4 questions.All previous questionnaires are valid and reliable instruments.

CONTACTS AND LOCATIONS:
Locations (1):
- Jazan Area Schools, Jizan, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No
After analysis of data, we will destroy all individual data to save participants privacy.

REFERENCES:
- [Derived] Alameer A, Mahfouz MS, Alamir Y, Ali N, Darraj A. Effect of Health Education on Female Teachers' Knowledge and Practices Regarding Early Breast Cancer Detection and Screening in the Jazan Area: a Quasi-Experimental Study. J Cancer Educ. 2019 Oct;34(5):865-870. doi: 10.1007/s13187-018-1386-9. PMID 29951902